CLINICAL TRIAL: NCT02398578
Title: Cystoscopic Ablation Via RF Energy Clinical Trial
Acronym: CARETI
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company closed May 1, 2019
Sponsor: Amphora Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1135-01
Record Dates: First submitted 2015-01-12; First posted 2015-03-25 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amphora OAB Device (Experimental): Specialized cystoscope that facilitates visualization and radiofrequency (RF) therapy for the treatment of OAB.
  Interventions: Device: Amphora OAB Device

INTERVENTIONS:
Device: Amphora OAB Device — Cystoscopic procedure to treat OAB

SUMMARY:
Phase I/II study to assess the safety and performance of the Amphora OAB system for treatment of urgency and frequency with or without urge incontinence caused by an overactive bladder.

DETAILED DESCRIPTION:
The study will enroll subjects with symptomatic idiopathic overactive bladder (OAB).

ELIGIBILITY:
Inclusion Criteria

Subjects must meet ALL the inclusion criteria to be eligible to participate in the study.

1. Non-pregnant, non-lactating female > 18 years old with a history of idiopathic OAB for ≥ 6 months
2. Have failed or are not a candidate for drug treatment
3. Subject is willing to provide Informed Consent, is geographically stable, understands the requirements for completing the bladder diary and is willing to comply with the required diary, follow up visits and testing schedules
4. Ambulatory without the aid of walking assistance a majority of the time (cane, walker etc.) and able to use toilet without assistance
5. Post-void residual (PVR) ≤ 100 ml NOTE: Subjects with a single PVR of >100 ml followed by two consecutive PVR measurements of ≤100 ml may be included in the study. The final acceptable PVR measurement will be recorded in the data.
6. Ability and willingness to self-catheterize in case this is necessary
7. 3 day Bladder Diary Criteria: Symptoms of OAB as evidenced by: Micturition frequency of ≥ 8 times/day And > 3 episodes of urgency urinary incontinence (UUI)

Exclusion Criteria

Subject will be excluded if ANY of the following conditions apply:

1. Planning on becoming pregnant during the 12 month study period
2. Current participation in any other conflicting interventional or OAB treatment study
3. Primary complaint of stress urinary incontinence or stress predominant mixed incontinence or functional incontinence
4. Any invasive or surgical intervention (e.g., radio frequency, implant, sling) involving the bladder, rectum or vaginal wall within the last 6 months
5. Ongoing complications of prior anti-incontinence surgery
6. Subject with 24-hour total urine volume voided greater than 3,000 ml as measured at screening period
7. Receiving electro-stimulation (e.g. PTNS or SNS) treatment within the last 15 days.

   NOTE: Subjects with an implanted SNS device that has not been active in the last 15 days is acceptable for enrollment
8. Botox treatment for OAB with 100u in the last 6 months OR Botox treatment with >100u in last 9 months
9. Urinary tract infection that is not resolved at the time of enrollment or had > 3 urinary tract infections (UTIs) within the last 12 months NOTE: If UTI is present at baseline screening, treatment with antibiotics and a negative urinalysis at least 7 days after the initial diagnosis of UTI will be acceptable for enrollment.
10. Documented spontaneous unprovoked urinary retention within the last 6 months
11. Anatomical conditions that would preclude the introduction and use of the device, in the opinion of the investigator, such as significant pelvic organ prolapse, urogenital prolapse visible at rest beyond the hymen, significant cystocele prolapse or high BMI
12. Current bleeding disorder or coagulopathies
13. Current use of antimuscarinics, β3 agonist or antispasmodics NOTE: subjects on these drugs must undergo a 2 week washout period prior to completing the baseline Bladder Diary.
14. Subject has been previously diagnosed with interstitial cystitis, bladder cancer or chronic pelvic pain syndrome.
15. Previous pelvic irradiation
16. Serum creatinine > twice the upper limit of normal within the last six months
17. Neurological disease affecting bladder function such as multiple sclerosis, spinal cord injuries, myasthenia gravis, Charcot-Marie-Tooth disease
18. Current hydronephrosis or hydroureter
19. Bladder outflow obstruction
20. Ureteral dysfunction, stricture or reflux

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Device-related complications through 24 month follow-up | 24 month

SECONDARY OUTCOMES:
Device Technical Success | During the study procedure
Procedural Success | During the study procedure
Change from Baseline of Quality of Life Scores | 4 weeks, 12 weeks, 6, 12, 18, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Roger Demochowski, MD, Principal Investigator — Vanderbilt University
Locations (4):
- Belgium (2):
  - University of Antwerp, Antwerp
  - University Hospital Ghent, Ghent
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Sherbrooke, Sherbrooke, Quebec